CLINICAL TRIAL: NCT00005711
Title: Intervention for Hispanic Children With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4920; R01HL045297 (NIH); HSC19900128H (Other: University of Texas Health Science Center San Antonio)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Control group children received routine medical care by their primary care providers as well as study visits every 6 months. At each study visit, following assessment of technique for using peak flow and metered dose inhalers, errors were corrected and children/families were coached on correct technique.
- Asthma self-management education (Experimental): Treatment group children and their families participated in the patient education program which consisted of four separate one-hour sessions. The topics were: symptoms of asthma, causes of asthma ("triggers"), medications, and peak flow. A bilingual nurse educator working one-on-one with the child and family members delivered these four sessions. The four sessions were delivered over a six week period. Culturally sensitive educational materials include both print (flip charts, take-home brochures) and videotape materials. The videotapes feature children from the clinic and highlight how they successfully manage their asthma. All materials are available in both English and Spanish.
  Interventions: Behavioral: Asthma self-management education

INTERVENTIONS:
Behavioral: Asthma self-management education — Treatment group children and their families participated in the patient education program which consisted of four separate one-hour sessions. The topics were: symptoms of asthma, causes of asthma ("triggers"), medications, and peak flow. A bilingual nurse educator working one-on-one with the child and family members delivered these four sessions. The four sessions were delivered over a six week period. Culturally sensitive educational materials include both print (flip charts, take-home brochures) and videotape materials. The videotapes feature children from the clinic and highlight how they successfully manage their asthma. All materials are available in both English and Spanish.
  Arms: Asthma self-management education

SUMMARY:
To design, implement, and evaluate an intervention program for Hispanic children with asthma which included both a physician education and a patient/family education component.

DETAILED DESCRIPTION:
BACKGROUND:

Although asthma affects 6-10 percent of children aged 6-16 years, the prevalence of asthma in Hispanic groups and the degree of resulting morbidity were unknown in 1990. The study sought to answer the following questions: 1) Would a physician education intervention result in improved medical management for Hispanic children with asthma who were cared for within the context of an outpatient clinic? 2) Would a focused educational intervention for Hispanic children with asthma and their families result in decreased morbidity and improved quality of life? If effective, the physician education and patient education programs could serve as models for the implementation of similar programs in outpatient clinic settings which serve Hispanic children with asthma.

The study was part of a demonstration and education initiative "Interventions for Control of Asthma Among Black and Hispanic Children" which was released by the NHLBI in June 1989.

DESIGN NARRATIVE:

Prior to enrollment of patients, all physicians participated in an intervention which included the following elements: a brief seminar about medical management for children with asthma, introduction of protocols in low chart format (algorithms), use of a standardized progress note from for children with asthma, a series of computer-based simulations and individualized feedback to physicians. The effectiveness of the physician education component in changing physician behavior was measured by pre- /post-test, chart audit, and performance on computer-based simulations.

One hundred sixty (160) Hispanic children with asthma, aged 6-15 years who were cared for in a pediatric residents' continuity clinic were enrolled for study. A research associate interviewed parents and children separately using standardized questionnaires to obtain information about 1) health beliefs, 2) reported health behavior, 3) knowledge and attitudes about asthma, 4) functional morbidity, 5) acculturation, and 6) socio-demographic factors. A research nurse performed spirometry on each subject. Additional information was obtained by review of medical records and school attendance records. Patients were then randomized into treatment and control groups. Treatment group patients and their families participated in the patient education intervention. The intervention consisted of a series of four videotapes and written materials which focused on major aspects of self-management for children with asthma. Patients and families received the four modules at one month intervals. Selected modules were reviewed with the research nurse at appointed visits approximately six, 9, and 12 months following enrollment. Follow-up data were obtained by interview, medical record review, and spirometry at six, 12, 18, and 24 months following enrollment.

Intervention and control group children were compared for morbidity (the number of emergency room visits, hospitalizations, school days missed) and quality of life (impact on family and functional status), after controlling for confounding variables. Secondary data analysis examined the effect of the intervention on knowledge, reported health behaviors, and post-intervention spirometry.

ELIGIBILITY:
Physician diagnosis of asthma; moderate severity (1997 criteria), ie. >= 2 ED visits or 1 hospitalization in past year or prescribed daily asthma medication.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 145 (Actual)
Dates: Start 1990-08; Primary Completion 2008-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Health care utilization | Enrollment, 12 months, 24 months
  ED visits; hospitalizations

SECONDARY OUTCOMES:
School absenteeism | Enrollment, 12 months, 24 months
  Number of school days misses per year
Lung function (FEV1 % predicted) | Enrollment, 6, 12, 18, 24 months
  FEV1 % predicted
Quality of life: Impact on Family | Enrollment, 6, 12, 18, 24 months
  Impact on Family scores
Quality of life: functional status | Enrollment, 6, 12, 18, 24 months
  functional impairment (FSII scores)
Self-management | Enrollment, 6, 12, 18, 24 months
  self-reported self-management behaviors

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hendricson WD, Wood PR, Hidalgo HA, Ramirez AG, Kromer ME, Selva M, Parcel G. Implementation of individualized patient education for Hispanic children with asthma. Patient Educ Couns. 1996 Nov;29(2):155-65. doi: 10.1016/0738-3991(96)00861-0. PMID 9006232
- [Result] Hendricson WD, Wood PR, Hidalgo HA, Kromer ME, Parcel GS, Ramirez AG. Implementation of a physician education intervention. The Childhood Asthma Project. Arch Pediatr Adolesc Med. 1994 Jun;148(6):595-601. doi: 10.1001/archpedi.1994.02170060049008. PMID 8193683
- [Result] Kromer ME, Prihoda TJ, Hidalgo HA, Wood PR. Assessing quality of life in Mexican-American children with asthma: impact-on-family and functional status. J Pediatr Psychol. 2000 Sep;25(6):415-26. doi: 10.1093/jpepsy/25.6.415. PMID 10980046
- [Result] Hidalgo H, Prihoda T, Arfken C, Evans D, Hanson J, Lapidus J, Malveaux F, Mellins R, Murphy S, Ramos C, Rand C, Strunk R, Sussman L, Thompson L, Wood P. Impact of home smoke exposure on black and hispanic children with asthma: a multi-center study. 1996. p. A420. (Am J Respir Crit Care Med; vol. 153).
- [Result] Wood PR, Hidalgo HA, Prihoda TJ, Kromer ME, Hendricson WD, Ramirez AG, Marinez YM. Asthma in hispanic children: a controlled study of the impact of patient education on morbidity. 1996. p. A276. (Am J Respir Crit Care Med; vol. 153).